CLINICAL TRIAL: NCT05608473
Title: The Effects of Video Based Cervical and Thoracal Posture Exercises on Head and Neck Posture, Muscular Endurance and Quality of Life in Office Workers
Brief Title: The Effects of Video Based Cervical and Thoracal Posture Exercises on Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İlke KARA, PT (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, İlke KARA, PT, Co-Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DEU-FTR-IK-02
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Physical Inactivity; Quality of Life
Keywords: Exercise; Posture; Workers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): A 10-minute video consisted of 14 exercises was uploaded to the computers of the participants in the exercise group. Participants were asked to do these exercises simultaneously with the video, 3 days in a week for 6 weeks. During theese weeks, the participants were checked by sms and they were asked to keep an exercise diary. For progression, the number of repetitions was increased in the 3rd week and the number of sets in the 5th week.
  Interventions: Other: Posture Exercises
- Control Group (No Intervention): The control group was given one session of training on postural correction.

INTERVENTIONS:
Other: Posture Exercises — A 10-minute video consisted of 14 cervical and thoracal postural exercises was uploaded to the computers of the participants. Participants were asked to do these exercises simultaneously with the video, 3 days in a week for 6 weeks. During theese weeks, the participants were checked by sms and they were asked to keep an exercise diary. For progression, the number of repetitions was increased in the 3rd week and the number of sets in the 5th week.
  Arms: Exercise Group

SUMMARY:
Aim of this study was investigate the effects of video-based cervical and thoracic postural exercises on muscle strength and endurance, hand grip strength, head-neck posture, quality of life and patient satisfaction in office workers.

DETAILED DESCRIPTION:
60 office workers between the ages of 25-65 were included in the study. Participants were randomly divided into Exercise group (EG, n=30) and Control group (KG, n=30). The video-based postural exercises were uploaded to the computers of the EG participants. They were asked to perform the exercises simultaneously with the video, 3 days a week for a total of 6 weeks. The control group was given one session of training on postural exercises. Cervical and scapular muscle strength and endurance, grip strength, craniovertebral angle, muscle endurance and strength, grip strength and head-neck posture measurements were made before the study and at the end of the 6th week. In addition, quality of life and satisfaction were evaluated with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* To be an office worker for at least 3 years
* To be literate

Exclusion Criteria:

* History of cervical, thoracic or shoulder surgeries
* Exercising regularly for the last 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Head-Neck Posture | Baseline
  Two markers were placed on the spinous process of C7 and targus of the ear. The angle was measured on the image taken with a digital camera.
Head-Neck Posture | At the end of the 6th week
  Two markers were placed on the spinous process of C7 and targus of the ear. The angle was measured on the image taken with a digital camera.
Muscle Strength | Baseline
  The cervical and scapular muscle strength was meausured with a Hand Held dynamometer (Lafayette Manual Muscle Test System™/ Model 01163-Lafayette Instrument Company, Lafayette, Indiana). Measurements were repeated three times, the average value was recorded.
Muscle Strength | At the end of the 6th week
  The cervical and scapular muscle strength was meausured with a Hand Held dynamometer (Lafayette Manual Muscle Test System™/ Model 01163-Lafayette Instrument Company, Lafayette, Indiana). Measurements were repeated three times, the average value was recorded.
Muscle Endurance | Baseline
  The muscular endurance of the deep cervical flexors was evaluated with the cranio-cervical flexion test. For general cervical flexor muscles, 0.5 kg weight was placed on the cervical region of the participant. The participant was asked to perform 10° cervical flexion while in cervical retraction, and the time he/she maintained this position was recorded. And for the trapezius and serratus anterior muscles, Scapular muscular endurance test was used.
Muscle Endurance | At the end of the 6th week
  The muscular endurance of the deep cervical flexors was evaluated with the cranio-cervical flexion test. For general cervical flexor muscles, 0.5 kg weight was placed on the cervical region of the participant. The participant was asked to perform 10° cervical flexion while in cervical retraction, and the time he/she maintained this position was recorded. And for the trapezius and serratus anterior muscles, Scapular muscular endurance test was used.
Handgrip Strength | Baseline
  Hand grip strength was assessed using a hand dynamometer (Jamar dynamometer / Promedics Ltd., Blackburn, Lancashire, UK) in a sitting position. The highest value from the three measurements was recorded.
Handgrip Strength | At the end of the 6th week
  Hand grip strength was assessed using a hand dynamometer (Jamar dynamometer / Promedics Ltd., Blackburn, Lancashire, UK) in a sitting position. The highest value from the three measurements was recorded.

SECONDARY OUTCOMES:
General Health | Baseline
  The QoL was assessed with the Short Form-36 QoL questionnaire administered under the supervision of the investigator. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). A score of zero indicates poor health, and a score of 100 indicates good health.
General Health | At the end of the 6th week
  The QoL was assessed with the Short Form-36 QoL questionnaire administered under the supervision of the investigator. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). A score of zero indicates poor health, and a score of 100 indicates good health.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal GELECEK, Professor, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No